CLINICAL TRIAL: NCT00016302
Title: The Use of Modified BFM +/- Compound 506U78 (Nelarabine) (NSC# 686673, IND #52611) in an Intensive Chemotherapy Regimen for the Treatment of T-Cell Leukemia
Brief Title: Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01857; COG-AALL00P2; U10CA098543 (NIH); CDR0000068620 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: T-cell Childhood Acute Lymphoblastic Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: interventions — Prednisone; Vincristine; Daunorubicin; Asparaginase; palmitoyl-L-asparaginase; Methotrexate; merphos; Cyclophosphamide; Cytarabine; Mercaptopurine; Leucovorin; Dexamethasone; Calcium Dobesilate; Doxorubicin; Thioguanine; Radiotherapy; Radiation; nelarabine; pegaspargase

ARMS (6):
- Regimen A (Experimental): See detailed description.
  Interventions: Drug: prednisone; Drug: vincristine sulfate; Drug: daunorubicin hydrochloride; Drug: asparaginase; Drug: methotrexate; Drug: cyclophosphamide; Drug: cytarabine; Drug: mercaptopurine; Drug: leucovorin calcium; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: thioguanine; Radiation: radiation therapy; Other: pharmacological study; Other: laboratory biomarker analysis
- Regimen B (Experimental): Induction (weeks 1-9): Patients receive treatment as in induction of regimen A.
  Consolidation (weeks 10-19): Patients receive treatment as in consolidation on regimen A.
  Reinduction (weeks 20-29): Patients receive treatment as in reinduction on regimen A and nelarabine IV on days 162-166.
  Maintenance (weeks 30-101): Patients receive oral mercaptopurine daily on days 1-28 and 36-56; oral methotrexate weekly; and nelarabine IV on days 29-33. Treatment repeats every 8 weeks for 4 courses. Beginning on week 62, patients receive vincristine IV once; oral prednisone three times daily for 5 days; oral mercaptopurine daily; and oral methotrexate weekly. Treatment repeats every 8 weeks for 5 courses.
  Interventions: Drug: prednisone; Drug: vincristine sulfate; Drug: daunorubicin hydrochloride; Drug: asparaginase; Drug: methotrexate; Drug: cyclophosphamide; Drug: cytarabine; Drug: mercaptopurine; Drug: leucovorin calcium; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: thioguanine; Radiation: radiation therapy; Drug: nelarabine; Other: pharmacological study; Other: laboratory biomarker analysis
- Regimen C (Experimental): Induction (weeks 1-5): Patients receive treatment as in induction (weeks 1-5) on regimen A and nelarabine IV over 1 hour on days 29-33.
  If bone marrow is M1, patients begin week 6 of induction therapy on day 36 or when peripheral blood counts recover. If bone marrow is M2, patients begin week 6 of induction therapy immediately. If bone marrow is M3, treatment discontinues.
  Induction (weeks 6-9): Patients receive treatment as in induction (weeks 6-9) on regimen A.
  Consolidation (weeks 10-19): Patients receive treatment as in consolidation on regimen A.
  Reinduction (weeks 20-29): Patients receive treatment as in reinduction on regimen B.
  Maintenance (weeks 30-101): Patients receive treatment as in maintenance on regimen B.
  Interventions: Drug: prednisone; Drug: vincristine sulfate; Drug: daunorubicin hydrochloride; Drug: asparaginase; Drug: methotrexate; Drug: cyclophosphamide; Drug: cytarabine; Drug: mercaptopurine; Drug: leucovorin calcium; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: thioguanine; Radiation: radiation therapy; Drug: nelarabine; Other: pharmacological study; Other: laboratory biomarker analysis
- Regimen D (Experimental): See detailed description.
  Interventions: Drug: prednisone; Drug: vincristine sulfate; Drug: daunorubicin hydrochloride; Drug: asparaginase; Drug: methotrexate; Drug: cyclophosphamide; Drug: cytarabine; Drug: mercaptopurine; Drug: leucovorin calcium; Drug: dexamethasone; Drug: thioguanine; Drug: nelarabine; Drug: pegaspargase; Radiation: radiation therapy; Other: pharmacological study; Other: laboratory biomarker analysis
- Regimen E (Experimental): Patients receive consolidation therapy, reinduction therapy, and maintenance therapy as in regimen D, but nelarabine is administered at a higher dose.
  Interventions: Drug: prednisone; Drug: vincristine sulfate; Drug: daunorubicin hydrochloride; Drug: asparaginase; Drug: methotrexate; Drug: cyclophosphamide; Drug: cytarabine; Drug: mercaptopurine; Drug: leucovorin calcium; Drug: dexamethasone; Drug: thioguanine; Drug: nelarabine; Drug: pegaspargase; Radiation: radiation therapy; Other: pharmacological study; Other: laboratory biomarker analysis
- Regimen F (Experimental): Patients receive nelarabine at a higher dose during induction therapy. Patients receive consolidation therapy, reinduction therapy, and maintenance therapy as in regimen E.
  Interventions: Drug: prednisone; Drug: vincristine sulfate; Drug: daunorubicin hydrochloride; Drug: asparaginase; Drug: methotrexate; Drug: cyclophosphamide; Drug: cytarabine; Drug: mercaptopurine; Drug: leucovorin calcium; Drug: dexamethasone; Drug: thioguanine; Drug: nelarabine; Drug: pegaspargase; Radiation: radiation therapy; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Drug: asparaginase — Given IM
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: methotrexate — Given IT and orally
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: cytarabine — Given IV or SC
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: mercaptopurine — Given orally
  Other Names: 6-mercaptopurine; 6-MP; Leukerin; MP
Drug: leucovorin calcium — Given IV or orally
  Other Names: CF; CFR; LV
Drug: dexamethasone — Given orally
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
  Arms: Regimen A; Regimen B; Regimen C
Drug: thioguanine — Given orally
  Other Names: 6-TG
Radiation: radiation therapy — Undergo cranial irradiation
  Other Names: irradiation; radiotherapy; therapy, radiation
  Arms: Regimen A; Regimen B; Regimen C
Drug: nelarabine — Given IV
  Other Names: 506U78; Arranon; GW506U78
  Arms: Regimen B; Regimen C; Regimen D; Regimen E; Regimen F
Drug: pegaspargase — Given IM
  Other Names: L-asparaginase with polyethylene glycol; Oncaspar; PEG-ASP; PEG-L-asparaginase
  Arms: Regimen D; Regimen E; Regimen F
Radiation: radiation therapy — Undergo craniocervical radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
  Arms: Regimen C; Regimen D; Regimen E; Regimen F
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. This phase II trial is studying several different combination chemotherapy regimens to see how well they work in treating patients with newly diagnosed acute lymphoblastic leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of the addition of nelarabine to modified multiagent Berlin-Frankfurt-Muenster-86 chemotherapy in patients with newly diagnosed T-cell acute lymphoblastic leukemia.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics and intracellular pharmacology of nelarabine in these patients.

OUTLINE: This is a pilot, multicenter study.

Prednisone Response Pre-Induction: All patients receive oral prednisone three times daily on days -7 to -1 and methotrexate intrathecally (IT) on day -7* of week 0. Good prednisone responders proceed to induction on regimen A. Poor prednisone responders proceed to induction on regimen C.

NOTE: *Patients who have received cytarabine IT within the week prior to study entry receive methotrexate IT on day -6.

Regimen A (good prednisone responders) (closed as of 2/27/03):

Induction (weeks 1-5): Patients receive vincristine IV on days 1, 8, and 15; oral prednisone three times daily on days 1-14; daunorubicin IV over 15 minutes on days 1, 8, 15, and 22; asparaginase intramuscularly (IM) on days 12, 15, 18, 22, 24, 27, 30, and 33; and methotrexate IT on day 1.

If bone marrow is M1, week 6 of induction therapy begins on day 36 or when peripheral blood counts recover. If bone marrow is M2, patients begin week 6 of induction therapy immediately. If bone marrow is M3, treatment discontinues. Those patients with minimal residual disease (MRD) on day 36 proceed to regimen B.

Induction (weeks 6-9): Patients receive cyclophosphamide IV over 1 hour on days 36 and 63; cytarabine IV over 72 hours on days 38-40, 45-47, 52-54, and 59-61; oral mercaptopurine daily on days 36-63; and methotrexate IT on days 45 and 59.

Consolidation (weeks 10-19): Patients receive oral mercaptopurine on days 64-119; methotrexate IV over 24 hours and leucovorin calcium IV, or orally as tolerated, on days 71, 85, 99, and 113; and methotrexate IT on days 71, 85, 99, and 113. (Patients begin methotrexate once blood counts recover and only if bone marrow is M1).

Reinduction (weeks 20-29): Patients receive oral dexamethasone three times daily on days 134-154; vincristine IV on days 141 and 148; doxorubicin IV over 15 minutes on days 134, 141, 148, and 155; and asparaginase IM on days 141, 144, 148, 151, 154, and 157. Beginning on day 169 or when blood counts recover, patients receive cyclophosphamide IV on day 169, cytarabine IV over 72 hours on days 171-173 and 178-180; oral thioguanine daily on days 169-182; and methotrexate IT on days 171 and 178. Patients also receive cranial irradiation for up to 10 days beginning on day 189.

Maintenance (weeks 30-101): Patients receive vincristine IV once; oral prednisone three times daily for 5 days; oral mercaptopurine daily; and oral methotrexate weekly. Treatment repeats every 8 weeks for 9 courses.

Regimen B (patients with MRD on day 36 of regimen A) (closed as of 2/27/03):

Induction (weeks 1-9): Patients receive treatment as in induction of regimen A.

Consolidation (weeks 10-19): Patients receive treatment as in consolidation on regimen A.

Reinduction (weeks 20-29): Patients receive treatment as in reinduction on regimen A and nelarabine IV on days 162-166.

Maintenance (weeks 30-101): Patients receive oral mercaptopurine daily on days 1-28 and 36-56; oral methotrexate weekly; and nelarabine IV on days 29-33. Treatment repeats every 8 weeks for 4 courses. Beginning on week 62, patients receive vincristine IV once; oral prednisone three times daily for 5 days; oral mercaptopurine daily; and oral methotrexate weekly. Treatment repeats every 8 weeks for 5 courses.

Regimen C (poor prednisone responders from stage 1 of study and all patients entered during stage 2 of study) (closed as of 2/27/03):

Induction (weeks 1-5): Patients receive treatment as in induction (weeks 1-5) on regimen A and nelarabine IV over 1 hour on days 29-33.

If bone marrow is M1, patients begin week 6 of induction therapy on day 36 or when peripheral blood counts recover. If bone marrow is M2, patients begin week 6 of induction therapy immediately. If bone marrow is M3, treatment discontinues.

Induction (weeks 6-9): Patients receive treatment as in induction (weeks 6-9) on regimen A.

Consolidation (weeks 10-19): Patients receive treatment as in consolidation on regimen A.

Reinduction (weeks 20-29): Patients receive treatment as in reinduction on regimen B.

Maintenance (weeks 30-101): Patients receive treatment as in maintenance on regimen B.

Regimen D (effective 5/2004):

Induction (weeks 1-5): Patients receive vincristine IV on days 1, 8, and 15; oral prednisone 3 times a day on days 1-14; daunorubicin IV over 15 minutes on days 1, 8, 15, and 22; nelarabine IV over 1 hour on days 29-33; asparaginase IM on days 12, 15, 18, 22, 24, 27, 30, and 33; and methotrexate IT on day 1.

If bone marrow is M1, week 6 of induction therapy begins on day 36 or when peripheral blood counts recover. If bone marrow is M2, patients begin week 6 of induction therapy immediately. If bone marrow is M3, treatment discontinues.

Induction (weeks 6-9): Patients receive cyclophosphamide IV over 1 hour on days 36 and 50; cytarabine IV or SC on days 36-39, 43-46, 50-53, and 57-60; oral mercaptopurine once daily on days 36-63; and methotrexate IT on days 43 and 57.

Patients who are poor responders to prednisone in induction therapy proceed to regimen F. Patients who are good responders to prednisone but have MRD after induction therapy proceed to regimen E. Patients who are good responders to prednisone and have no MRD after induction therapy continue therapy on regimen D.

Consolidation (weeks 10-19): Patients must have M1 marrow to proceed. Patients receive oral mercaptopurine on days 70-126; methotrexate IV over 24 hours on days 77, 84, 91, and 98; leucovorin calcium IV or orally every 6 hours on days 78-79, 85-86, 92-93, and 99-100; and methotrexate IT on days 77, 84, 91, and 98.

Reinduction (weeks 20-29): Patients < 13 years old receive dexamethasone 3 times daily on days 140-161. Patients ≥ 13 years old receive oral dexamethasone on days 140-146 and 155-161; nelarabine IV on days 169-173; vincristine IV over 15 minutes on days 140, 147, and 153; pegaspargase IM on day 143; cyclophosphamide IV on day 176; cytarabine IV or SC on days 176-179 and 183-186; oral thioguanine on days 176-189; and methotrexate IT on days 176 and 183. Patients with CNS disease undergo craniocervical radiotherapy beginning on day 196 and continuing for 7-10 days.

Maintenance (weeks 30-61): Patients receive oral mercaptopurine on days 1-28 and 36-56; oral methotrexate on days 1, 8, 15, 22, 36, 43, and 50; and nelarabine IV on days 29-33. Treatment repeats every 8 weeks for 4 courses.

Maintenance (weeks 62-101): Patients receive vincristine IV on day 1; oral dexamethasone twice daily on days 1-5; oral mercaptopurine on days 1-56; and oral methotrexate on days 1, 8, 15, 22, 29, 36, 43, and 50. Treatment repeats every 8 weeks for 5 courses.

Regimen E (good responders to induction prednisone but with MRD) (effective 5/2004): Patients receive consolidation therapy, reinduction therapy, and maintenance therapy as in regimen D, but nelarabine is administered at a higher dose.

Regimen F (poor responders to induction prednisone) (effective 5/2004): Patients receive nelarabine at a higher dose during induction therapy. Patients receive consolidation therapy, reinduction therapy, and maintenance therapy as in regimen E.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 100 patients (30 for regimens A, B, and C; 70 for regimens D, E, and F) will be accrued for this study within 9-29 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed T-cell acute lymphoblastic leukemia with greater than 25%bone marrow blasts (M3)

  * High-risk disease, defined as meeting at least 1 of the following criteria:

    * WBC at least 50,000/mm^3
    * Age 10 years or over
* Patients with WBC at least 25,000/mm^3 AND at least 50% peripheral blood blasts are eligible provided bone marrow aspiration was contraindicated (e.g., patient was not eligible for anesthesia or sedation due to respiratory distress secondary to anterior mediastinal mass)
* Concurrent registration to POG 9900 within the past 8 days required
* Performance status - Karnofsky 50-100% (over 10 years of age)
* Performance status - Lansky 50-100% (10 years of age and under)
* See Disease Characteristics
* Bilirubin no greater than 1.5 mg/dL
* SGPT less than 5 times normal
* Creatinine normal
* Creatinine clearance or glomerular filtration rate at least 60 mL/min
* No pre-existing neuropathy of grade 2 or worse unless due to leukemic infiltration
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior biologic therapy
* No more than 72 hours since prior intrathecal cytarabine
* No other prior chemotherapy
* Prior steroids allowed
* No chronic steroid treatment for another disease
* Prior emergency radiotherapy to mediastinum for severe respiratory distress allowed

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2001-04; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Grade 3+ unusual CNS toxicities assessed using NCI CTCAE v. 3.0 | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Dunsmore, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States